CLINICAL TRIAL: NCT06355856
Title: Phase IV, National, Unicentric, Comparative, Double-Blind, Randomized, Non- Inferiority Clinical Trial to Evaluate the Efficacy and Safety of DNN.22.17.036 Compared to 10573048700 in the Treatment of Androgenetic Alopecia
Brief Title: Efficacy/ Safety of DNN.22.17.036 in Male Patients With Pattern Hair Loss
Acronym: CAPELLI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-PNT-04(01/22)
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNN.22.17.036 (Experimental): Apply 1 ml to the bald area of the scalp, twice a day for 180 days.
  Interventions: Drug: DNN.22.17.036
- 10573048700 (Active Comparator): Apply 1 ml to the bald area of the scalp, twice a day for 180 days.
  Interventions: Drug: 10573048700

INTERVENTIONS:
Drug: DNN.22.17.036 — Apply twice daily to the affected area and around it.
  Arms: DNN.22.17.036
Drug: 10573048700 — Apply twice daily to the affected area and around it.
  Arms: 10573048700

SUMMARY:
Evaluation of the efficacy and safety of DNN.22.17.036 versus 10573048700 in the treatment of male pattern hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and consent to participate in this clinical research, expressed by signing the Informed Consent Form (ICF)
* Male participants age 25 or older and 60 age or younger
* Participants who have an intact scalp in the area of product analysis
* Participants with androgenetic alopecia (AGA) with AGA Norwood-Hamilton Scale > II
* Participants with at least 20% telogen effluvium of evaluated by Tricholab

Exclusion Criteria:

* Participants who have used immunosuppressants in the 3 months prior to signing the ICF
* Participants with other causes of hair loss or scalp dermatoses
* Participants who have received hair loss treatment in the last 6 months
* Participants with uncontrolled medical conditions, kidney and liver disease
* Participants with a history of hair transplantation, malignancy, hematologic disorders, thyroid dysfunction, malnutrition, and other dermatologic disorders that contribute to hair loss

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentage variation of hairs in the hair loss phase | 180 days
  Percentage variation of hairs in the hair loss phase (telogen hairs), by image analysis with the FotoFinder Leviacam®, after 180 days of treatment.

IPD SHARING:
Plan to Share IPD: No